CLINICAL TRIAL: NCT06683339
Title: Assessment of Functional Capacity in Children with Chronic Kidney Disease
Brief Title: Functional Capacity in Children with Chronic Kidney Disease
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2022/04-27
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Disease(CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with chronic kidney disease

SUMMARY:
The aim of our study is to assess the functional capacity of children with chronic kidney disease using various tests.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with chronic kidney disease
* Being clinically stable
* Being between 6-18 years old
* Volunteering to participate in the research

Exclusion Criteria:

* Having a musculoskelatal disease that may affect functional capacity measurement
* Having a cognitive problem

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with chronic kidney disease will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | 1st day
  Exercise capacity will be evaluated with 6 minute walk test.
Exercise capacity | 1st day
  Exercise capacity will be assessed using 2 minute walk test
Exercise capacity | 1st day
  Exercise capacity will be assessed using 3 minute step test.

SECONDARY OUTCOMES:
Muscle strength | 1st day
  Knee extensor and hand grip strength will be measured using a hand dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Firat, Principal Investigator — Kirsehir Ahi Evran University; Naciye Vardar-Yagli, Study Director — Hacettepe University; Bora Gulhan, Study Chair — Hacettepe University; Melda Saglam, Study Chair — Hacettepe University; Aydan Asli Aksel-Uylar, Study Chair — Hacettepe University; Rezan Topaloglu, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)